CLINICAL TRIAL: NCT00996788
Title: Anti Free Radical & Anti Inflammatory Effect & Safety of Rebamipide in Chronic Gastritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PT Otsuka Indonesia (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 037-IOB-0701
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Dyspepsia; Chronic Gastritis
Keywords: Patients suffering of dyspepsia due to chronic gastritis
MeSH Terms: conditions — Dyspepsia | interventions — rebamipide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rebamipide (Experimental): Rebamipide 100 mg tid for 28 days
  Interventions: Drug: Rebamipide

INTERVENTIONS:
Drug: Rebamipide — Rebamipide 100 mg tid for 28 days

SUMMARY:
To study the anti free radical & inflammatory effect and safety of Rebamipide in patients suffering of dyspepsia due to chronic gastritis.

ELIGIBILITY:
Inclusion Criteria:

Patients who

1. are 18 - 80 years old
2. have symptoms of dyspepsia that need endoscopic examination
3. are suffering from chronic moderate to severe gastritis which is confirmed endoscopically
4. are able to give informed concern

Exclusion Criteria:

Patients who

1. are treated with drugs that induce gastritis/ulcer, such as: NSAID
2. are chronic alcoholism,
3. are drug abuser
4. are contraindicated for endoscopy examination
5. has erosive or ulcerative esophagitis
6. has peptic ulcer that has been confirmed by endoscopy
7. has pyloric stenosis
8. has active gastrointestinal bleeding
9. has major absorption disorder
10. has history of gastric surgery
11. with renal disorder (creatinine > 2 mg/dL)
12. with liver disease ( SGOT, SGPT, bilirubin)
13. have hematologic disorder ( confirmed with hemoglobin, erythrocytes, leucocytes,differential blood count)
14. are suffering from congestive gastropathy due cirrhosis
15. are suffering from congestive heart disease
16. are pregnant or giving breast feeding
17. are hypersensitive to Rebamipide
18. are treated with gastroprotective drugs such as : teprenone, sucralfate.
19. are treated with acid suppressing medicine (H2A, PPI)
20. are treated with antibiotics, mesalazine (Salofalk)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of Rebamipide 100 mg t.i.d. in reducing gastric mucosal damage due to free radical and inflammation | 2 times (at day-0 and day-28)

SECONDARY OUTCOMES:
To confirm the improvement of dyspepsia syndrome | 3 times (at day-0, day-7 and day-28)

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Rani, MD, Principal Investigator — Division of Gastroenterology Department of Internal Medicine - Cipto Mangunkusumo Hospital, Faculty of Medicine University of Indonesia
Locations (1):
- Division of Gastroenterology Department of Internal Medicine - Cipto Mangunkusumo Hospital, Faculty of Medicine University of Indonesia, Jakarta, Indonesia